CLINICAL TRIAL: NCT07034209
Title: An Open-label, Single-arm, Multicenter Clinical Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetic Characteristics, and Immunogenicity of Plonmarlimab in Subjects With Rheumatic and Immunological Disease-associated Haemophagocytic Lymphohistiocytosis (HLH) (Also Known as Macrophage Activation Syndrome (MAS))
Brief Title: A Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetic Characteristics, and Immunogenicity of Plonmarlimab in Subjects With Rheumatic and Immunological Disease-associated Haemophagocytic Lymphohistiocytosis (HLH) (Also Known as Macrophage Activation Syndrome (MAS))
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TJ Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THZ0103-201
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Hemophagocytic Lymphohistiocytoses
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — plonmarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plonmarlimab (Experimental)
  Interventions: Drug: Plonmarlimab

INTERVENTIONS:
Drug: Plonmarlimab — Subjects receive Plonmarlimab 6 mg/kg or 10 mg/kg, administered intravenously, once weekly for 8 weeks.

SUMMARY:
This study adopts an open-label, single-arm, multicenter design to evaluate the efficacy, safety, tolerability, immunogenicity, and PK characteristics of Plonmarlimab administration in patients with rheumatic and immunological disease-associated HLH (MAS), and to explore biomarkers related to the efficacy of Plonmarlimab.

ELIGIBILITY:
Inclusion Criteria:

1. Age: This study will include subjects aged 16 to 80 years (inclusive), of any gender.
2. The subject is willing to participate in this study and voluntarily signs the informed consent form. For minor subjects aged 16 years (inclusive) to less than 18 years, written informed consent must be signed by both the subject and the subject's legal guardian
3. Diagnosed with haemophagocytic lymphohistiocytosis (HLH) according to the HLH-2004 diagnostic criteria (see Appendix 1 for details. HLH-2004 diagnostic criteria)，
4. Diagnosed with a rheumatic and immunological disease,including:Systemic juvenile idiopathic arthritis (sJIA);Adult Onset Still's Disease (AOSD);Systemic lupus erythematosus (SLE)
5. The subject (including the subject's partner) has no plans for pregnancy from the screening period until 28 days after the last dose and is willing to use contraceptive measures (oral oestrogens, oestrogens, vaginal rings, etc., cannot be used; see Appendix 5. Contraceptive Measures, Definition of Women of Childbearing Potential, and Contraception Requirements for acceptable contraceptive measures).

Exclusion Criteria:

1. Known pathogenic gene mutation or abnormal perforin expression and CD107a degranulation assay indicating primary haemophagocytic lymphohistiocytosis, or a family history of primary haemophagocytic lymphohistiocytosis.
2. Subjects who:

   1. Are receiving tumour necrosis factor (TNF) antagonists (anti-TNF), interleukin-1 (IL-1) antagonists [anti-IL-1, e.g., canakinumab, anakinra], Janus kinase inhibitors (JAKi), or interleukin-6 (IL-6) antagonists [anti-IL-6, e.g., tocilizumab] at the time of initiating Plonmarlimab treatment;
   2. Received Etoposide (VP-16) for MAS treatment within 7 days before the first dose;
   3. Increased the dose or type of non-biologic agents (e.g., immunosuppressants, immunomodulators, antimalarials) for the treatment of rheumatic and immunological diseases within 3 days before the first dose. Unless the investigator determines it is expected to be ineffective and it is discontinued before the first dose. Specific drugs for immunosuppressants, immunomodulators.
3. History of allergy to any component of the investigational drug.
4. Lung disorder: Including but not limited to asthma, chronic obstructive pulmonary disease (COPD), interstitial lung disease, alveolar proteinosis, pulmonary granulomatosis, etc., AND abnormal pulmonary function tests: forced vital capacity (FVC) <80% of predicted value, or FEV1/FVC <70%, etc.; or cases where the investigator's comprehensive assessment indicates that the subject has a pre-existing lung disorder significantly affecting pulmonary function and is unsuitable for participation in this clinical study.
5. Cardiovascular disorder: History of acute myocardial infarction or unstable angina pectoris, severe arrhythmia (e.g., multifocal frequent premature ventricular contractions, ventricular tachycardia, ventricular fibrillation) within the last 6 months; New York Heart Association (NYHA) functional classification III-IV (see Appendix 6. NYHA Functional Classification).
6. History of neoplasm malignant within the past 5 years (whether treated or not), with the exception of successfully treated cutaneous basal cell or squamous cell carcinoma.
7. Other diseases: Subjects currently have clinically significant and clinically unstable or uncontrolled acute or chronic disease (e.g., acute pneumonia, pulmonary arterial hypertension, diabetic ketoacidosis, pancreatitis acute, etc.), or planned medical/surgery procedures; or place the subject at undue risk, or affect the subject's ability to voluntarily participate in the study.
8. Infection: Subjects with investigator-assessed uncontrolled infection during the screening period.
9. Subjects with Mycobacterium tuberculosis infection, including those with latent infection positive by "T-SPOT" or "QuantiFERON" test.
10. Positive for any of the following: hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab), treponema pallidum antibody test. If hepatitis B core antibody (HBcAb) test is positive, an additional hepatitis B DNA (HBV-DNA) test will be performed; subjects with HBV-DNA above the lower limit of detection will be excluded.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate,ORR | At the end of Week 8

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Renji Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Beijing Peking Union Medical College Hospital, Beijing
  - Beijing Peking University People's Hospital, Beijing
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Ruijin Hospital Of Shanghai Jiao tong University School of Medicine, Shanghai